CLINICAL TRIAL: NCT04357938
Title: Risk Stratification With Chest Computed Tomography to Rule-out Suspected SARS-CoV-2 Infections of Unspecific Symptomatic Patients Before Hospital Admission
Brief Title: Risk Stratification With Chest CT to Rule-out Suspected SARS-CoV-2 Infections
Acronym: SCout
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Ulf Teichgräber, Professor of Radiology, Chairman of Radiology Dep., Jena University Hospital
Other Study IDs: IDIR-001-2020
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: interventions — Postmortem Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CT-imaging — Chest CT to rule out pneumonia in PCR negative, nonspecific symptomatic patients to prevent the spread of SARS-CoV-2 within the hospital.
  Other Names: Chest computed tomography

SUMMARY:
The study objective is to investigate the diagnostic value and consistency of chest CT as compared with comparison to RT-PCR assay in COVID-19 in patients which were stratified for hospital admission.

DETAILED DESCRIPTION:
To prevent spreading of the new coronavirus (SARS-CoV-2) from patients who are infected but in whom infection was not detected by means of Reverse transcription polymerase chain reaction (RT-PCR) and who are to be admitted to ordinary wards of hospitals, we aimed to determine validity of exclusion of pneumonia immediately before admission by means of chest computed tomography.

Patients admitted to the emergency department of the university hospital Jena with Covid-19 symptoms (temperature > 37.5°C; respiratory and/or gastrointestinal symptoms) whose RT-PCR test resulted negative, undergo a chest CT scan. Those patients without pulmonary infiltrates can be safely ruled out for Covid-19. Thus, CT has perfect selectivity evidence regarding pulmonary infiltrates; it has limited selectivity concerning the pathogenesis of the infiltration.

The study objective is to investigate the diagnostic value and consistency of chest CT as compared with comparison to RT-PCR assay in COVID-19 in patients which were stratified for hospital admission.

The hypothesis is that chest CT has the greatest clinical evidence (no detection of lung infiltration) when the RT-PCT is tested negative. We assume that chest CT has a high sensitivity for diagnosis of respiratory dominant COVID-19. A pulmonary COVID-19 in epidemic areas can be best ruled out when chest CT is negative for the presence of infiltrations of the lung parenchyma. This is described by the SNOUT principle which is an acronym for 'Sensitive test when Negative rules OUT the disease' under the condition of a low pretest probability.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Provided written informed consent
* Intended hospital admission for any reason
* Symptoms that suggest infection with SARS-CoV-2
* Participant agrees to rt PCR and antibody test (SARS-CoV-2)

Exclusion Criteria:

* < 18 years
* Pregnancy cannot be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unspecific symptoms of SARS-CoV-2 infection who are to be admitted to hospital for any disease and who provide written informed consent to undergo rt-PCR, chest CT, and antibody test.
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of chest CT in detecting pneumonia in unspecific symptomatic patients who are to be admitted to hospital and who are rt-PCR negative for SARS-CoV-2. | At hospital admission
  Positive likelihood ratio (LR+) Negative likelihood ratio (LR-)

SECONDARY OUTCOMES:
Sensitivity and specificity of chest CT in patients with pulmonary comorbidities | At hospital admission
  Sensitivity and specificity of chest CT in detecting pneumonia in unspecific symptomatic patients with pulmonary comorbidities who are to be admitted to hospital and who are rt-PCR negative for SARS-CoV-2.
Sensitivity and specificity of chest CT in patients with cardiovascular comorbidities | At hospital admission
  Sensitivity and specificity of chest CT in detecting pneumonia in unspecific symptomatic patients with cardiovascular comorbidities who are to be admitted to hospital and who are rt-PCR negative for SARS-CoV-2.
Sensitivity and specificity of chest CT in patients with malignancy | At hospital admission
  Sensitivity and specificity of chest CT in detecting pneumonia in unspecific symptomatic patients with malignancy who are to be admitted to hospital and who are rt-PCR negative for infection with SARS-CoV-2.
Sensitivity and specificity of chest CT in patients with immunodeficiency | At hospital admission
  Sensitivity and specificity of chest CT in detecting pneumonia in unspecific symptomatic patients with immunodeficiency who are to be admitted to hospital and who are rt-PCR negative for SARS-CoV-2.

OTHER OUTCOMES:
Predictive value of specific chest CT findings for detection of SARS-CoV-2 | At hospital admission
  Predictive value of chest CT

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Teichgräber, Prof. Dr., Principal Investigator — Department of Radiology, Jena University Hospital, Germany
Locations (1):
- Jena University Hospital, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Teichgraber U, Malouhi A, Ingwersen M, Neumann R, Reljic M, Deinhardt-Emmer S, Loffler B, Behringer W, Lewejohann JC, Stallmach A, Reuken P. Ruling out COVID-19 by chest CT at emergency admission when prevalence is low: the prospective, observational SCOUT study. Respir Res. 2021 Jan 12;22(1):13. doi: 10.1186/s12931-020-01611-w. PMID 33435973